CLINICAL TRIAL: NCT01188421
Title: Medications Development for Drug Abuse Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-018125; NA_00037871 (Other: JHUSOM IRB); R01DA018125 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-08-11; First posted 2010-08-25 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Opioid Related Disorders; Opioid Dependence; Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Clonidine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- buprenorphine (Active Comparator): Sublingual buprenorphine/naloxone tablets (or placebo)
  Interventions: Drug: Buprenorphine/naloxone
- clonidine (Active Comparator): Oral clonidine tablets (or placebo)
  Interventions: Drug: Clonidine
- tramadol ER (Experimental): Oral tramadol tablets (or placebo)
  Interventions: Drug: Tramadol ER

INTERVENTIONS:
Drug: Buprenorphine/naloxone — up to 8/2 mg Sublingual (SL) per day
  Other Names: Suboxone
  Arms: buprenorphine
Drug: Clonidine — up to 0.8 mg per day (oral)
  Other Names: Catapres
  Arms: clonidine
Drug: Tramadol ER — up to 600 mg per day
  Other Names: Ultram
  Arms: tramadol ER

SUMMARY:
This is a study of tramadol as an agent for short-term opioid withdrawal treatment. A randomized, double blind clinical trial comparing the efficacy and safety of tramadol to clonidine and buprenorphine in the short-term treatment of opioid withdrawal will be conducted. Opioid dependent participants will be treated on a residential unit. The primary outcome measure is opioid withdrawal symptoms.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Participants in this study will be males and females between the ages of 18 and 60 years.
* Applicants must be opioid dependent based upon the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) (SCID); in addition, they must have an opioid positive urine during the screening process (or have evidence of opioid withdrawal).
* They must be healthy, with no significant medical illnesses (e.g., insulin dependent diabetes), and without significant psychiatric illness (e.g., schizophrenia) besides their drug dependence.
* Females will have a pregnancy test prior to study enrollment, and if found to be pregnant will be excluded and referred to a substance abuse program for pregnant women (the Center for Addiction and Pregnancy) on the campus.
* Volunteers will also be excluded if they have pre-admission hypotension (due to the use of clonidine in the study).
* Applicants with a history of seizures (including substance-related seizures, such as alcohol withdrawal related) will be excluded.
* Alcohol and/or sedative dependence will be specific exclusionary criteria (given the small risk of seizures associated with tramadol use).
* Allergies to any of the study medications will be grounds for exclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Dunn KE, Tompkins DA, Bigelow GE, Strain EC. Efficacy of Tramadol Extended-Release for Opioid Withdrawal: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):885-893. doi: 10.1001/jamapsychiatry.2017.1838. PMID 28700791

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine: Sublingual buprenorphine/naloxone tablets (or placebo)
  Buprenorphine/naloxone: up to 8/2 mg SL per day
Period: Overall Study
Arm/Group | Buprenorphine | Tramadol ER | Clonidine
Started | 31 | 36 | 36
Completed | 28 | 26 | 22
Not Completed | 3 | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Tramadol ER | Clonidine | Total
Number analyzed (Participants) | 31 | 36 | 36 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.9) | 40.9 (9.7) | 41.5 (10.5) | 41.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 15
  Male | 27 | 31 | 30 | 88
Race/Ethnicity, Customized [Number; unit: percentage of participants]
  Caucasian | 38.7 | 47.2 | 41.6 | 42.5

OUTCOME MEASURES:

1. Primary Outcome: Mean Ratings on Clinical Opiate Withdrawal Scale (COWS) Measure of Withdrawal During Double-blind Taper (7-days) and Post-taper (7-days) Period.
Description: Outcomes represent mean peak withdrawal as rated on the Clinical Opiate Withdrawal Scale (COWS) total score. Withdrawal was collected 7 times daily and daily peak values were identified for each participant and averaged together as a function of group. Primary outcomes were mean peak results from the 7-day taper period and first 7 days post-taper. The COWS is an 11-item observer-rated measure of opioid withdrawal severity. Items are rated on individual Likert scales and the total score range is 0-47. Higher values indicate more severe withdrawal.
Time Frame: 14 days total
Population: Repeated measures ANOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Buprenorphine | Tramadol ER | Clonidine
Number analyzed (Participants) | 31 | 36 | 36
units on a scale
  Taper Day 1 | 7.79 (1.68) | 8.41 (0.70) | 8.28 (0.71)
  Taper Day 2 | 6.16 (2.03) | 6.10 (0.72) | 8.00 (0.46)
  Taper Day 3 | 4.76 (1.77) | 3.77 (0.35) | 5.85 (0.66)
  Taper Day 4 | 4.21 (1.77) | 4.25 (0.52) | 4.70 (0.57)
  Taper Day 5 | 4.31 (2.11) | 3.25 (0.37) | 3.32 (0.41)
  Taper Day 6 | 4.06 (1.63) | 3.39 (0.45) | 3.57 (0.57)
  Taper Day 7 | 3.51 (1.28) | 3.69 (0.53) | 3.86 (0.64)
  Post Taper Day 1 | 4.82 (1.62) | 3.36 (0.44) | 3.27 (0.37)
  Post Taper Day 2 | 5.62 (1.90) | 4.48 (0.60) | 4.09 (0.60)
  Post Taper Day 3 | 6.23 (1.75) | 3.28 (0.28) | 3.68 (0.38)
  Post Taper Day 4 | 5.49 (1.66) | 3.13 (0.24) | 3.82 (0.46)
  Post Taper Day 5 | 5.87 (1.69) | 2.75 (0.24) | 3.27 (0.35)
  Post Taper Day 6 | 4.91 (1.62) | 2.57 (0.26) | 2.91 (0.31)
  Post Taper Day 7 | 4.91 (1.69) | 2.30 (0.23) | 2.41 (0.31)
Statistical Analysis 1: Comparison: Buprenorphine vs Tramadol ER vs Clonidine; A power analysis determined 40 participants in each group would detect a moderate effect size, assuming an alpha of 0.05 and 80% power. Due to the expiration of buprenorphine tablets, recruitment was terminated after enrolling 103 participants. This study utilized an Intent-to-Treat (ITT) analysis. The ITT analysis includes all volunteers who signed informed consent, were randomized into the study's treatment conditions, and took at least 1 dose of study medication; Test type: Superiority; p = .275, ANOVA — Main effect of Group (e.g., Buprenorphine, Tramadol, Clonidine) on COWS Total Score Ratings; F-value for main effect of Group = 1.310
Statistical Analysis 2: Comparison: Buprenorphine vs Tramadol ER vs Clonidine; Test type: Superiority; p = 0.03, ANOVA — Main effect for Phase (e.g., Stabilization, Taper, Post-Taper) on COWS total score; F-value for main effect of Phase = 3.570
Statistical Analysis 3: Comparison: Buprenorphine vs Tramadol ER vs Clonidine; Test type: Superiority; p = 0.092, ANOVA — Main effect for Group x Phase interaction on COWS Total Score; F-value for the main effect of Group x P = 2.030

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the Taper and Post-Taper periods (approximately 18-19 days). No Adverse Events reported from Stabilization phase (7-10 day period) since this occurred prior to primary experimental manipulation and randomization to study drug (clonidine, tramadol, buprenorphine).
Description: Standard terminology
Arm/Group | Buprenorphine | Tramadol ER | Clonidine
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 28/31 | 31/36 | 32/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (N=31) | Tramadol ER (N=36) | Clonidine (N=36)
Chills (General disorders) | 9 (11) | 13 (20) | 17 (21)
Drowsiness (General disorders) | 1 (1) | 1 (1) | 4 (4)
Headache (General disorders) | 17 (22) | 14 (22) | 10 (19)
Lethargy (General disorders) | 2 (2) | 1 (1) | 3 (4) — stupor or coma from disease
Malaise (General disorders) | 2 (2) | 1 (1) | 2 (2) — uneasiness or indisposition
Abdominal Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 6 (7)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 6 (10) | 8 (11) | 9 (9) — High heart rate
Abdominal Cramp (Gastrointestinal disorders) | 9 (9) | 4 (4) | 14 (16)
Diarrhea (Gastrointestinal disorders) | 13 (18) | 9 (15) | 20 (25)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 9 (11) | 4 (6)
Flatulance (Gastrointestinal disorders) | 2 (2) | 4 (5) | 3 (3)
Indigestion (Gastrointestinal disorders) | 2 (2) | 4 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 9 (10)
Vomitting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5) | 5 (6) — pain in joint
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (9) | 2 (2)
Cramp Lower Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle Ache (Musculoskeletal and connective tissue disorders) | 11 (14) | 11 (16) | 10 (10)
Pain Lower Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 2 (2)
Agitation (Nervous system disorders) | 2 (2) | 1 (1) | 4 (4)
Anxiety (Nervous system disorders) | 8 (9) | 10 (15) | 10 (11)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Fatigue (Nervous system disorders) | 2 (2) | 6 (7) | 5 (10)
Insomnia (Nervous system disorders) | 12 (18) | 15 (18) | 14 (17)
Irritability (Nervous system disorders) | 3 (3) | 9 (13) | 12 (12)
Restlessness (Nervous system disorders) | 12 (15) | 15 (20) | 11 (11)
Shaky (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 10 (13) | 9 (14) | 8 (8)
Cough (General disorders) | 0 (0) | 0 (0) | 2 (2) — non-productive
Nasal Congestion (General disorders) | 5 (6) | 5 (5) | 6 (7)
Rhinitis (General disorders) | 0 (0) | 4 (5) | 2 (2)
Rhinorrhea (General disorders) | 13 (15) | 10 (14) | 10 (16)
Yawning (General disorders) | 8 (11) | 4 (4) | 6 (6) — Excessively
Piloerection (General disorders) | 5 (6) | 4 (4) | 1 (1)
Sweat Increased (General disorders) | 6 (8) | 5 (6) | 6 (6)
Hot Flashes (Eye disorders) | 6 (7) | 7 (7) | 8 (9)
Lacrimation Increased (Eye disorders) | 2 (2) | 8 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes